CLINICAL TRIAL: NCT04322864
Title: Web-based Instrument Intervention for Individuals with Shoulder Pain: Randomized Controlled Trial
Brief Title: Web-based Instrument Intervention for Individuals with Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Vander Gava, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eHealthRCT
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain; Musculoskeletal Diseases
MeSH Terms: conditions — Shoulder Pain; Musculoskeletal Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-person supervised intervention (Active Comparator)
  Interventions: Other: Therapeutic exercises
- Web-based instrument intervention (Experimental)
  Interventions: Other: Therapeutic exercises

INTERVENTIONS:
Other: Therapeutic exercises — Patients will perform strengthening exercises focusing on scapulothoracic muscles and shoulder lateral rotators.

SUMMARY:
Introduction: Shoulder pain is a condition of high prevalence in the general population. Studies indicate that physiotherapeutic treatment with exercise is effective in reducing pain and restoring function in patients with shoulder pain. Patients may have difficulty accessing the physiotherapy service due to the cost of treatment, transportation to the service, and long waiting lines. A possible solution is the use of a web-based exercise prescription instrument to increase access to physiotherapy for shoulder pain patients. Objective: To verify the effects of an intervention with a web-based instrument compared to a in person and supervised intervention. Methods: This study is a controlled, randomized, blinded clinical trial. There will be 184 individuals with shoulder pain who will be randomly assigned to two groups. One group will receive a web-based instrument intervention and the other group will receive the in person and supervised intervention. The intervention will consist of strengthening exercises with emphasis on the lateral rotator and scapulothoracic muscles. The primary outcome will be pain and disability (SPADI, Shoulder Pain and Disability Index), and the secondary outcomes will be function (DASH questionnaire, Disabilities of the Arm, Shoulder and Hand), self-efficacy (CPSS, Chronic Pain Self-Efficacy Scale), kinesiophobia (Cover Scale), patient expectation of treatment (7-point Likert Scale), and patient satisfaction (Global Change Assessment Scale). All outcomes will be measured before and after 12 weeks of treatment (2x/week), after 6 months and 12 months from the end of treatment. Normality of data will be verified by Kolmogorov Smirnov's test. Differences between groups will be verified using the mixed linear models with the interaction terms versus time. The effect size will be calculated for the variables between the groups. The significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60;
* Self-reported pain of intensity equal to or greater than 3 points on the numerical pain scale (NDT) at rest or arm movement in the anterolateral region of the shoulder;
* Duration of at least 3 months of shoulder pain;
* Have a mobile phone with Android 4.1 or higher.

Exclusion Criteria:

* History of trauma related to the onset of symptoms;
* History of clavicle, scapula or humerus fracture;
* History of surgical stabilization or rotator cuff repair;
* History of shoulder dislocation;
* Pain related to the cervical spine;
* Adhesive capsulitis;
* Systemic disease involving the joints and cognitive alteration that makes it impossible to carry out questionnaires or use the mobile application.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline Shoulder Pain and Disability to 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Pre (baseline) treatment, post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Shoulder Pain and Disability will be measured with Shoulder Pain and Disability Index with scores ranging from 0 to 100 (higher score reflects higher pain and disability)

SECONDARY OUTCOMES:
Change in baseline Pain to 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Pre (baseline) treatment, post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Pain will be measured with 11 point - Numerical Rating Pain Scale with scores ranging from 0 (no pain) to 10 (maximum pain).
Change in baseline Function to 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Pre (baseline) treatment, post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Function will be measured with Disabilities of the Arm, Shoulder and Hand with scores ranging from 0 to 100 (higher score reflects higher disability)
Change in baseline Self-efficacy to 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Pre (baseline) treatment, post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Self-efficacy will be measured with Chronic Pain Self-Efficacy Scale with scores ranging from 30 to 300 (higher score reflects greater self-efficacy)
Change in baseline Kinesiophobia to 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Pre (baseline) treatment, post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Kinesiophobia will be measured with Tampa Scale of Kinesiophobia with scores ranging from 17 to 68 (higher score reflects higher kinesiophobia)
Patients' expectation with the treatment at baseline | Pre (baseline) treatment
  Patients' expectation with the treatment will be measured with a 7-point Likert scale ranging from 1 (worse than ever) to 7 (totally recovered).
Patients' Self-perception of improvement with the treatment at 12 weeks, 6 months (follow-up 1) and 12 months (follow-up 2) | Post treatment (12 weeks), after 6 months (follow-up 1) and 12 months (follow-up 2)
  Self-perception of improvement will be measured with the Global Rating of Change Scale with scores ranging from -7 to +7 (A higher score indicates higher recovery from the condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
At the end of the clinical trial will be published the Study Protocol and Statistical Analysis Plan (SAP), if any researcher wants more information can request. The Informed Consent Form (ICF) can also be available.